CLINICAL TRIAL: NCT02205671
Title: Building Better Caregivers: Development and Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Kate Lorig, Professor Emeritus, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 29894
Record Dates: First submitted 2014-07-29; First posted 2014-07-31 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Providing Care for People With Memory Problems
Keywords: caregiving; chronic illness; patient education; self management
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Building Better Caregivers Small-group Workshop
  Interventions: Behavioral: Building Better Caregivers Small-group Workshop

INTERVENTIONS:
Behavioral: Building Better Caregivers Small-group Workshop

SUMMARY:
The program consists of a 6-week small-group workshop for caregivers of people with memory problems.

The goal of the study is to evaluate in a one year longitudinal study, program effectiveness in reducing caregiver stress, depression, fatigue, burden, days lost from work and improving sleep, healthful behaviors and self-efficacy

DETAILED DESCRIPTION:
The Building Better Caregivers workshop meets for 2.5 hours per week for 6 weeks in small groups of 10-16. It is peer-led (leaders already trained in the Stanford model must take a 2-day cross-training before leading a BBC workshop).

Participants will learn self-management skills such as decision making, goal setting, action planning, stress management, dealing with difficult behaviors, working with the health care system, planning for the future,building an exercise program, communication skills, healthy eating, etc.

All participants will complete follow up questionnaires and 6 and 12 months. They will have the option of completing the questionnaire by mail or telephone interview.

Once a particular workshop site is identified by a partner organization, Stanford will provide packets of consents and questionnaires to the site coordinator(non-Stanford). The site coordinator will either schedule an extra hour for the first meeting of the 6-week series, or an orientation meeting held a week or so before the workshop begins. During this time, the coordinator will announce to the prospective subjects that this study is being conducted and that they are invited to participate, and will pass out a consent, questionnaire and consent copy to each prospective participant. The consent and questionnaire are self-administered.

This study is longitudinal, so no randomization will take place.

Stanford holds no meetings, but receives the data. The site coordinators hold the orientation meetings. The workshops are scheduled by the various organizations, and they determine when and how the orientation time is scheduled. It will vary from site to site.

ELIGIBILITY:
Inclusion Criteria:

* Family or friend caregiver of someone with cognitive impairment for at least 10 hours per week
* 18 years of age or older
* Able to attend a workshop 2.5 hours per week for 6 weeks
* Speaks English

Exclusion Criteria:

* Professional caregiver
* Under 18 years of age
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Fatigue | baseline-1 year
  visual numeric 0-10 scale
Pain | baseline-1 year
  visual numeric 0-10 scale
stress | baseline-1 year
  visual numeric 0-10 scale
problems sleeping | baseline-1 year
  visual numeric 0-10 scale
depression (PHQ-8) | baseline-1 year
  8 item 0-3 scale
self-efficacy for caregiving | baseline-1 year
  9-item 1-10 scale
caregiver stress | baseline-1 year
  13-item 3 point scale
caregiver burden | baseline-1 year
  12-item 5 point scale
health care utilization (doctor, emergency department, hospital) | baseline-1 year
  number of times/days in past 6 month visited doctor, emergency department, hospital
exercise | baseline- 1 year
  number of minutes of exercise in past week
general health | baseline-1 year
  single item scale of overall health

SECONDARY OUTCOMES:
care partner health utilization | baseline- 1 year
  number of MD ER hospital visits for person being cared for in past 6 months
carepartners general health | baseline-1 year
  single item scale of overall health of person being cared for

CONTACTS AND LOCATIONS:
Overall Officials: Kate Lorig, DRPH, Principal Investigator — Stanford School of Medicine
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States